CLINICAL TRIAL: NCT02232698
Title: Randomised Controlled Study to Evaluate the Impact of Novel Glucose Sensing Technology on Hypoglycaemia in Type 1 Diabetes
Brief Title: An Evaluation of Novel Glucose Sensing Technology on Hypoglycaemia in Type 1 Diabetes (IMPACT)
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ADC-CI-APO-13019
Record Dates: First submitted 2014-09-03; First posted 2014-09-05 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-02

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Sensing Technology; Type 1 Diabetes,
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sensor Based Glucose Monitoring System (Experimental): Standard sensing system use for 6 months.
  Interventions: Device: Sensor Based Glucose Monitoring System
- Standard Blood Glucose Monitoring (Active Comparator): Subjects randomised to the control group will be given blood glucose meters for monitoring for the 6 months study duration.
  Interventions: Device: Standard Blood Glucose Monitoring

INTERVENTIONS:
Device: Sensor Based Glucose Monitoring System — Subjects will wear the Abbott Sensor Based Glucose Monitoring System (unmasked) for 6 months to monitor their glucose levels.
  All subjects will wear a masked Abbott Sensor Based Glucose Monitoring System, for 14 days prior to randomisation (Sensor glucose measurements not visible during this time).
  Arms: Sensor Based Glucose Monitoring System
Device: Standard Blood Glucose Monitoring — Subjects will use an Abbott Blood Glucose Monitoring System (standard blood glucose meter) for 6 months to monitor their glucose levels. A 14-day masked wear of the Abbott Sensor Based Glucose Monitoring System is included for these subjects at the 3 and 6 month time point, to collect glycaemic variability data for comparison to the intervention group of the study (Sensor glucose measurements not visible during this time).
  All subjects will wear a masked Abbott Sensor Based Glucose Monitoring System, for 14 days prior to randomisation (Sensor glucose measurements not visible during this time).
  Arms: Standard Blood Glucose Monitoring

SUMMARY:
The purpose of this study is to evaluate the impact of the Abbott Sensor Based Glucose Monitoring System on hypoglycaemia compared to Self Monitoring Blood Glucose (SMBG) testing using a randomised controlled study design in adults with Type 1 diabetes using insulin.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Type 1 diabetes for ≥ 5 years
2. On their current insulin regimen for ≥ 3 months prior to study entry
3. Screening HbA1c result ≤ 7.5% (58 mmol/mol)
4. Reports self testing of blood glucose levels on a regular basis equivalent to a minimum of 3 times daily for at least 2 months prior to study entry
5. In the investigator's opinion the subject is considered technically capable of using the Abbott Sensor Based Glucose Monitoring System
6. Aged 18 years or over.

Exclusion Criteria:

1. Subject has been diagnosed with hypoglycaemic unawareness (i.e. subject has a diagnosis of impaired awareness of hypoglycaemia recorded in their medical notes OR in the investigator's opinion the subject currently experiences less than minimal warning symptoms for impending hypoglycaemia)
2. Subject is currently prescribed animal insulin
3. Subject is currently prescribed oral steroid therapy or is likely to require oral steroid therapy for any acute or chronic condition during the study
4. Has known allergy to medical grade adhesives
5. Currently participating in another device or drug study that could affect glucose measurements or glucose management
6. Currently using a Continuous Glucose Monitoring (CGM) device or has used one within the previous 4 months
7. Currently using Sensor augmented pump therapy
8. Is planning to use a CGM device at any time during the study
9. A female subject who is pregnant or planning to become pregnant within the study duration
10. A breast feeding mother
11. Currently receiving dialysis treatment or planning to receive dialysis during the study
12. Has a pacemaker
13. Has experienced an acute myocardial infarction within previous 6 months
14. Has a concomitant disease or condition that may compromise subject safety including; unstable coronary heart disease, cystic fibrosis, serious psychiatric disorder, or any other uncontrolled medical condition
15. Has experienced an episode of confirmed or suspected diabetic ketoacidosis (DKA) in the previous 6 months
16. In the investigator's opinion, the subject is considered unsuitable for inclusion in the study for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2014-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Matthaei, Principal Investigator — Diabetes Center Quakenbruck
Locations (23):
- Austria (6):
  - VIVIT-Institut am Akad. Lehrkrankenhaus Feldkirch, Innere Medizin und Kardiologie, Feldkirch
  - Medizinische Universität Graz Abteilung für Innere Medizin, Klin. Abteilung für Endokrinologie und Stoffwechsel, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - Diakonissen-Krankenhaus Salzburg, Salzburg
  - Klinik fuer Innere Medizin III Medizinische Universitaet Wien, Vienna
  - Wilhelminenspital Medzin 5, Vienna
- Germany (5):
  - Diabetes Klinik Bad Mergentheim, Bad Mergentheim
  - Zentrum für Diabetologie Hamburg Bergedorf, Hamburg
  - Diabetes-Zentrum Hannover-Nord, Hanover
  - Diabetes Center Quakenbruck, Quakenbrück
  - Versdias GmbH, Sūlzbach-Rosenberg
- Netherlands (6):
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Onze Lieve Vrouwe gasthuis ( OLVG), Amsterdam
  - Amphia Ziekenhuis, Breda
  - Bethesda Diabetes Research Center, Hoogeveen
  - Medisch Centrum Haaglanden, The Hague
  - St. Antonius Ziekenhuis, Utrecht
- Spain (3):
  - Hospital Germans Trias i Pujol, Badalona
  - Clinica Diabetologica, Gijón
  - Servicio de Endocrinología Hospital Unversitario Cruces, Vizcaya
- Sweden (3):
  - Falu Lasarett, Falun
  - Karolinska Universitetssjukhuset Solna, Solna
  - Karolinska Universitetssjukhuset Huddinge, Stockholm

REFERENCES:
- [Derived] Oskarsson P, Antuna R, Geelhoed-Duijvestijn P, Krӧger J, Weitgasser R, Bolinder J. Impact of flash glucose monitoring on hypoglycaemia in adults with type 1 diabetes managed with multiple daily injection therapy: a pre-specified subgroup analysis of the IMPACT randomised controlled trial. Diabetologia. 2018 Mar;61(3):539-550. doi: 10.1007/s00125-017-4527-5. Epub 2017 Dec 23. PMID 29273897
- [Derived] Rayman G, Kroger J, Bolinder J. Could FreeStyle Libre sensor glucose data support decisions for safe driving? Diabet Med. 2018 Apr;35(4):491-494. doi: 10.1111/dme.13515. Epub 2017 Oct 14. PMID 28945936
- [Derived] Bolinder J, Antuna R, Geelhoed-Duijvestijn P, Kroger J, Weitgasser R. Novel glucose-sensing technology and hypoglycaemia in type 1 diabetes: a multicentre, non-masked, randomised controlled trial. Lancet. 2016 Nov 5;388(10057):2254-2263. doi: 10.1016/S0140-6736(16)31535-5. Epub 2016 Sep 12. PMID 27634581

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 328 subjects consented and enrolled into the study. Eighty-seven (87) of these failed screening or withdrew before randomisation. Two hundred and forty-one (241) subjects were randomised and 211 completed the study.
Groups:
- Sensor Based Glucose Monitoring System: Standard sensing system use for 6 months.
  Sensor Based Glucose Monitoring System: Subjects will wear the Abbott Sensor Based Glucose Monitoring System (unmasked) for 6 months to monitor their glucose levels.
  All subjects will wear a masked Abbott Sensor Based Glucose Monitoring System, for 14 days prior to randomisation (Sensor glucose measurements not visible during this time).
- Standard Blood Glucose Monitoring: Subjects randomised to the control group will be given blood glucose meters for monitoring for the 6 months study duration.
  Standard Blood Glucose Monitoring: Subjects will use an Abbott Blood Glucose Monitoring System (standard blood glucose meter) for 6 months to monitor their glucose levels. A 14-day masked wear of the Abbott Sensor Based Glucose Monitoring System is included for these subjects at the 3 and 6 month time point, to collect glycaemic variability data for comparison to the intervention group of the study (Sensor glucose measurements not visible during this time).
  All subjects will wear a masked Abbott Sensor Based Glucose Monitoring System, for 14 days prior to randomisation (Sensor glucose measurements not visible during this time).
Period: Overall Study
Arm/Group | Sensor Based Glucose Monitoring System | Standard Blood Glucose Monitoring
Started | 120 | 121
Completed | 110 | 101
Not Completed | 10 | 20
Not completed — Pregnancy | 1 | 1
Not completed — Met exclusion criteria | 1 | 1
Not completed — Had device-associated symptoms | 7 | 0
Not completed — Non-compliance with study device | 1 | 4
Not completed — Allocated to control group | 0 | 3
Not completed — Withdrawal by Subject | 0 | 11

BASELINE CHARACTERISTICS:
Population: 2 pregnant subjects (1 in each group) were excluded from all efficacy analysis (as stated in the protocol).
Groups:
- Total: Total of all reporting groups
Arm/Group | Sensor Based Glucose Monitoring System | Standard Blood Glucose Monitoring | Total
Number analyzed (Participants) | 119 | 120 | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (13.1) | 45.0 (14.6) | 43.7 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 61 | 103
  Male | 77 | 59 | 136
Screening HbA1c [Mean (Standard Deviation); unit: %] | 6.73 (0.52) | 6.74 (0.59) | 6.74 (0.56)
Screening HbA1c [Mean (Standard Deviation); unit: mmol/mol] | 50.1 (5.7) | 50.2 (6.5) | 50.1 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Time Spent <70 mg/dL
Description: Difference in time <70 mg/dL between intervention and control group assessed in days 194 to 208 adjusting for baseline (days 1 to 15).
Time Frame: Baseline and Days 194 to 208
Population: 1 subject from the standard blood glucose monitoring group had no baseline sensor data and could not be included in the analysis of sensor data.
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Sensor Based Glucose Monitoring System | Standard Blood Glucose Monitoring
Number analyzed (Participants) | 119 | 119
hours per day
  Baseline | 3.38 (2.31) | 3.44 (2.62)
  Days 194-208 | 2.03 (1.93) | 3.27 (2.58)
Statistical Analysis 1: Comparison: Sensor Based Glucose Monitoring System vs Standard Blood Glucose Monitoring; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -1.24, Standard Error of Mean 0.239

2. Secondary Outcome: HbA1c at 6 Months
Description: Difference in HbA1c between intervention and control group at day 208 adjusting for baseline HbA1c at day 1
Time Frame: Baseline and Day 208
Measure: Mean (Standard Deviation); unit: percentage of Glycated Haemoglobin
Arm/Group | Sensor Based Glucose Monitoring System | Standard Blood Glucose Monitoring
Number analyzed (Participants) | 119 | 120
percentage of Glycated Haemoglobin
  Baseline | 6.79 (0.52) | 6.78 (0.64)
  Day 208 | 6.94 (0.65) | 6.95 (0.66)
Statistical Analysis 1: Comparison: Sensor Based Glucose Monitoring System vs Standard Blood Glucose Monitoring; Test type: Superiority or Other; p = 0.9556, ANCOVA; Mean Difference (Final Values) = 0.00, Standard Error of Mean 0.059

3. Secondary Outcome: Time Spent <55 mg/dL and <40 mg/dL
Description: Difference in time <55 mg/dL & <40 mg/dL (hours per day) between intervention and control group assessed in days 194 to 208 adjusting for baseline (days 1 to 15).
Time Frame: Baseline and Days 194 to 208
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Sensor Based Glucose Monitoring System | Standard Blood Glucose Monitoring
Number analyzed (Participants) | 119 | 119
hours per day
  Time spent <55 mg/dL, Baseline | 1.59 (1.42) | 1.77 (1.86)
  Time spent <55 mg/dL, Days 194-208 | 0.80 (0.96) | 1.65 (1.97)
  Time spent <40 mg/dL, Baseline | 0.59 (0.85) | 0.75 (1.11)
  Time spent <40 mg/dL, Days 194-208 | 0.26 (0.47) | 0.73 (1.41)
Statistical Analysis 1: Comparison: Sensor Based Glucose Monitoring System vs Standard Blood Glucose Monitoring; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical analysis of time spent <55 mg/dL; Mean Difference (Final Values) = -0.82, Standard Error of Mean 0.175
Statistical Analysis 2: Comparison: Sensor Based Glucose Monitoring System vs Standard Blood Glucose Monitoring; Test type: Superiority or Other; p = 0.0003, ANCOVA — Statistical analysis of time spent <40 mg/dL; Mean Difference (Final Values) = -0.46, Standard Error of Mean 0.122

4. Secondary Outcome: Frequency of Episodes <70 mg/dL, <55 mg/dL and <40 mg/dL
Description: Difference in frequency of episodes <70 mg/dL, <55 mg/dL and <40 mg/dL (number per day) between intervention and control group assessed in days 194 to 208 adjusting for baseline (days 1 to 15).
Time Frame: Baseline and Days 194-208
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of episodes per day
Arm/Group | Sensor Based Glucose Monitoring System | Standard Blood Glucose Monitoring
Number analyzed (Participants) | 119 | 119
number of episodes per day
  Frequency of episodes <70 mg/dL, Baseline | 1.81 (0.90) | 1.67 (0.80)
  Frequency of episodes <70 mg/dL, Days 194-208 | 1.32 (0.81) | 1.69 (0.83)
  Frequency of episodes <55 mg/dL, Baseline | 0.96 (0.65) | 0.92 (0.73)
  Frequency of episodes <55 mg/dL, Days 194-208 | 0.56 (0.55) | 0.92 (0.74)
  Frequency of episodes <40 mg/dL, Baseline | 0.39 (0.43) | 0.44 (0.51)
  Frequency of episodes <40 mg/dL, Days 194-208 | 0.19 (0.29) | 0.43 (0.55)
Statistical Analysis 1: Comparison: Sensor Based Glucose Monitoring System vs Standard Blood Glucose Monitoring; Statistical analysis of frequency of episodes <70 mg/dL; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.45, Standard Error of Mean 0.089
Statistical Analysis 2: Comparison: Sensor Based Glucose Monitoring System vs Standard Blood Glucose Monitoring; Statistical analysis of frequency of episodes <55 mg/dL; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.38, Standard Error of Mean 0.074
Statistical Analysis 3: Comparison: Sensor Based Glucose Monitoring System vs Standard Blood Glucose Monitoring; Statistical analysis of frequency of episodes <40 mg/dL; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.22, Standard Error of Mean 0.050

5. Secondary Outcome: Time Spent >180 mg/dL and >240 mg/dL
Description: Difference in time >180 mg/dL and >240 mg/dL (hours per day) between intervention and control group assessed in days 194 to 208 adjusting for baseline (days 1 to 15).
Time Frame: Baseline and Days 194 to 208
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Sensor Based Glucose Monitoring System | Standard Blood Glucose Monitoring
Number analyzed (Participants) | 119 | 119
hours per day
  Time spent >180 mg/dL, Baseline | 5.62 (2.48) | 5.80 (3.11)
  Time spent >180 mg/dL, Days 194-208 | 6.16 (3.05) | 6.08 (3.20)
  Time spent >240 mg/dL, Baseline | 1.85 (1.44) | 1.91 (1.70)
  Time spent >240 mg/dL, Days 194-208 | 1.67 (1.36) | 2.06 (1.61)
Statistical Analysis 1: Comparison: Sensor Based Glucose Monitoring System vs Standard Blood Glucose Monitoring; Statistical analysis of time spent >180 mg/dL; Test type: Superiority or Other; p = 0.5623, ANCOVA; Mean Difference (Final Values) = 0.19, Standard Error of Mean 0.329
Statistical Analysis 2: Comparison: Sensor Based Glucose Monitoring System vs Standard Blood Glucose Monitoring; Statistical analysis for time spent >240 mg/dL; Test type: Superiority or Other; p = 0.0247, ANCOVA; Mean Difference (Final Values) = -0.37, Standard Error of Mean 0.163

6. Secondary Outcome: Time in Range
Description: Difference in time in range 70-180 mg/dL between intervention and control group assessed in days 194 to 208 adjusting for baseline (days 1 to 15 time in range).
Time Frame: Baseline and Days 194 to 208
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Sensor Based Glucose Monitoring System | Standard Blood Glucose Monitoring
Number analyzed (Participants) | 119 | 119
hours per day
  Baseline | 15.0 (2.5) | 14.8 (2.8)
  Days 194-208 | 15.8 (2.9) | 14.6 (2.9)
Statistical Analysis 1: Comparison: Sensor Based Glucose Monitoring System vs Standard Blood Glucose Monitoring; Test type: Superiority or Other; p = 0.0006, ANCOVA; Mean Difference (Final Values) = 1.0, Standard Error of Mean 0.30

7. Secondary Outcome: Number of Glucose Measurements Performed
Description: Number of blood glucose fingerstick tests per day by intervention and control group during baseline (days 1 to 15) and days 194 to 208. The number of sensor scans performed performed by the intervention group during days 15 to 208.
Time Frame: Days 1 to 208
Measure: Mean (Standard Deviation); unit: number of measurements per day
Arm/Group | Sensor Based Glucose Monitoring System | Standard Blood Glucose Monitoring
Number analyzed (Participants) | 106 | 93
number of measurements per day
  Number of fingerstick tests, Baseline | 5.5 (2.0) | 5.8 (1.7)
  Number of fingerstick tests, Days 194-208 | 0.6 (1.0) | 5.6 (2.2)
  Number of sensor scans, Days 15-208 | 15.1 (6.9) | NA (NA) — Number of sensor scans does not apply to this group as they did not use the sensor to self-manage their glucose levels.

8. Secondary Outcome: System Utilisation
Description: System utilisation assessed by percentage of sensor glucose data collected by the intervention group
Time Frame: Days 15 to 208
Population: 112 subjects included in the analysis, 7 were not included due to missing data.
Measure: Mean (Standard Deviation); unit: percentage of sensor glucose collected
Arm/Group | Sensor Based Glucose Monitoring System
Number analyzed (Participants) | 112
percentage of sensor glucose collected | 92.8 (7.3)

9. Secondary Outcome: Change in Diabetes Treatment Satisfaction Questionnaire (DTSQc) Scores From Day 1 to Day 208
Description: The Diabetes Treatment Satisfaction Questionnaire change (DTSQc) score is used to assess relative change in participant satisfaction from baseline. The questionnaire consists of 8 items, 6 of which (1 and 4 through 8) assess treatment satisfaction. Each item is rated on a 7-point Likert scale (which ranges from -3 (much less satisfied) to +3 (much more satisfied). The scores from the 6 treatment satisfaction items are summed to a Total Treatment Satisfaction Score, which ranges from -18 (much less satisfied) to +18 (much more satisfied).
  There is one question to assess the change in perceived frequency of Hypoglycaemia and one question to assess change in perceived frequency of Hyperglycaemia. Each question is rated on a 7-point Likert scale (-3 to +3), -3 (much less of the time now) to +3 (much more of the time now).
  The ANCOVA adjusts for baseline DTSQs (status version).
Time Frame: Baseline and Day 208
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sensor Based Glucose Monitoring System | Standard Blood Glucose Monitoring
Number analyzed (Participants) | 103 | 86
units on a scale
  Hyperglycaemia | -0.6 (1.6) | 0.5 (1.2)
  Hypoglycaemia | -0.3 (1.6) | 0.1 (1.1)
  Treatment Satisfaction | 13.4 (5.5) | 7.2 (6.2)
Statistical Analysis 1: Comparison: Sensor Based Glucose Monitoring System vs Standard Blood Glucose Monitoring; Statistical analysis of perceived frequency of hyperglycaemia; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -1.0, Standard Error of Mean 0.22
Statistical Analysis 2: Comparison: Sensor Based Glucose Monitoring System vs Standard Blood Glucose Monitoring; Statistical analysis of perceived frequency of hypoglycaemia; Test type: Superiority or Other; p = 0.0713, ANCOVA; Mean Difference (Final Values) = -0.4, Standard Error of Mean 0.22
Statistical Analysis 3: Comparison: Sensor Based Glucose Monitoring System vs Standard Blood Glucose Monitoring; Statistical analysis of total treatment satisfaction score; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 6.1, Standard Error of Mean 0.84

ADVERSE EVENTS:
Time Frame: Adverse events collected from enrolment (6 months)
Description: In addition to the serious adverse events listed below, 1 subject reported a serious adverse event of hypoglycaemia during the baseline phase (prior to randomisation), this subject was subsequently randomised to the Sensor Based Glucose Monitoring group.
  No serious adverse events were related to the study device.
Arm/Group | Sensor Based Glucose Monitoring System | Standard Blood Glucose Monitoring
Serious Adverse Events (participants affected / at risk) | 4/120 | 4/121
Other Adverse Events (participants affected / at risk) | 33/120 | 24/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sensor Based Glucose Monitoring System (N=120) | Standard Blood Glucose Monitoring (N=121)
atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sensor Based Glucose Monitoring System (N=120) | Standard Blood Glucose Monitoring (N=121)
medical device site reaction (General disorders) | 10 (13) | 0 (0)
influenza (Infections and infestations) | 7 (7) | 7 (7)
nasopharyngitis (Infections and infestations) | 19 (20) | 17 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days